CLINICAL TRIAL: NCT01199120
Title: Cognitive Effects of Omega-3 Supplements in Children With Mild to Moderate Malnutrition
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad Autonoma de Ciudad Juarez (Other)
Responsible Party: Veronica Portillo Reyes - PI, Universidad Autonoma de Ciudad Juarez
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UACJ-ICSA-VPortillo-01
Record Dates: First submitted 2010-09-06; First posted 2010-09-10 (Estimated); Last update posted 2010-09-10 (Estimated); Status verified 2010-09

CONDITIONS: Malnourishment
Keywords: Omega-3; Cognition; Malnourishment
MeSH Terms: conditions — Malnutrition | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omega 3 (Experimental)
  Interventions: Dietary Supplement: Omega 3

INTERVENTIONS:
Dietary Supplement: Omega 3 — measure of efficacy of omega-3 fatty acids supplement on cognition and academic performance in children attending elementary school.

SUMMARY:
Adequate nutrition is one of the critical biological processes to learning and cognitive development of children. And is understandable that malnourishment affect these processes. Moreover, in recent decades it has been investigated the beneficial effects of Omega-3 in cognitive development and academic performance. However, studies have been limited. Therefore is of interest to know the effects that has supplement with Omega-3 for children 8-12 years with malnutrition in a randomized, blind, placebo-controlled.

DETAILED DESCRIPTION:
Adequate nutrition is one of the most critical biological processes to learning and cognitive development of children, and malnourishment is understandable these processes are affected. Moreover, in recent decades is has been investigated the beneficial effects of Omega-3 in cognitive development and academic performance. However, studies have been limited. The present study will investigate the efficacy of omega-3 fatty acids supplement on cognition and academic performance in children attending elementary school.

The study will follow a randomized, double-blind, placebo-controlled design in which children aged 6-12 years will followed for a period of three months to assess cognitive development, academic performance and nutritional status . Intervention will take place in elementary schools, where children will receive two intervention products daily and one more in their houses. The products will contain omega-3 fatty acids, placebo, or only neuropsychological evaluation (control group with normal nutrition children). At baseline, and 3months cognitive tests will be administered and assess nutritional status. Compliance will be measured weekly.

We hypothesize that after 12 months of intervention, children consuming omega-3 fatty acids will have statistically significant higher improvement in scores on cognitive tests, than placebo and normal nutrition children.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 8- 12 years that attending the selected elementary schools.
2. Whit no problems for swallowing pills.
3. Willing to participate in the study and perform all measurements including anthropometry and cognitive evaluation
4. Informed consent signed by parent or caregiver.
5. Parents intend to stay in the study for three months.

Exclusion Criteria:

1. Neurological and/or hormonal illnesses.
2. Children using medication which interferes with study measurements.
3. Omega-3 or any other vitamin supplements consumption within the last 6 months.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2009-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Cognitive development and performance | three months
  Comparation of the effects of parallels treatment

SECONDARY OUTCOMES:
Size effect of intervention | three months

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Autonoma de Ciudad Juarez, Juárez, Chihuahua, Mexico

REFERENCES:
- [Derived] Portillo-Reyes V, Perez-Garcia M, Loya-Mendez Y, Puente AE. Clinical significance of neuropsychological improvement after supplementation with omega-3 in 8-12 years old malnourished Mexican children: a randomized, double-blind, placebo and treatment clinical trial. Res Dev Disabil. 2014 Apr;35(4):861-70. doi: 10.1016/j.ridd.2014.01.013. Epub 2014 Feb 6. PMID 24508294